CLINICAL TRIAL: NCT04662554
Title: Pilot Study of a 1-Millimeter Resolution Clinical PET System in Head and Neck Cancer Imaging
Brief Title: Study of a 1-Millimeter Resolution Clinical Positron Emission Tomography (PET) System in Head and Neck Cancer Imaging
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Goldman Sachs Foundation (Unknown); Wallace H. Coulter Foundation (Other); Emerson Collective (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB-55884; ENT0080 (Other: OnCore)
Record Dates: First submitted 2020-11-06; First posted 2020-12-10 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Novel PET Camera (Experimental): Patients already undergoing a PET/CT scan for HNC will afterwards undergo a PET scan with the proposed device, thus no additional radioactivity is needed as part of this study.
  Interventions: Device: 1-mm Resolution Clinical PET camera

INTERVENTIONS:
Device: 1-mm Resolution Clinical PET camera — 1-Millimeter Resolution Clinical PET System in Head and Neck Cancer (HNC) Imaging

SUMMARY:
The purpose of this study is to gain initial experience imaging HNC patient using a new PET camera, a 1mm spacial resolution. The goal is to understand image quality of the system and to see how it works in a clinical environment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE(S): Gain initial experience imaging head/neck cancer patients using a novel PET camera comprising two opposing panels with 1 millimeter spatial resolution.

SECONDARY OBJECTIVE(S):

1. Determine the radioactive dose and scan time required for this novel 1 millimeter (mm) resolution clinical PET camera.
2. Images obtained with the 1 mm resolution PET camera will be compared to conventional PET imaging (which will serve as gold standard) for image quality and lesion/node visualization.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-confirmed diagnosis of HNC
2. Patient scheduled to undergo surgery for HNC
3. Scheduled to have a PET/CT study on a conventional PET/CT system
4. Age greater than or equal to 19 years of age.

Exclusion Criteria:

1. Additional condition, or extenuating circumstance that, in the opinion of the investigator, may interfere with study compliance.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Acquiring PET images of HNC patients with the 1 mm resolution PET imaging device. | Day 1
  PET images of HNC patients with the 1 mm resolution PET imaging device will be qualitatively accessed whether the camera can visualize the primary lesion, including heterogeneity and lymph nodes will be assessed.

SECONDARY OUTCOMES:
Measure image quality of the 1 mm resolution PET imaging device | Day 1
  Image quality of the 1 mm resolution PET imaging device (scale 1-5) with 5 being highest 'image quality' will be assessed to understand radioactive dose and scan time required for a given desired image quality.

CONTACTS AND LOCATIONS:
Overall Officials: Eben Rosenthal, Ph.D, Principal Investigator — Stanford Universiy
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No